CLINICAL TRIAL: NCT06649877
Title: A Randomized Clinical Study to Evaluate the Impact of Injection Site (Thigh vs Abdomen) on the Pharmacokinetics and Relative Bioavailability of Subcutaneously Injected MK-6194 in Healthy Adult Participants
Brief Title: MK-6194 Site of Injection Study in Healthy Adult Participants (MK-6194-013)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 6194-013; MK-6194-013 (Other: MSD)
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abdomen Injection (Experimental): Participants will receive a single dose of MK-6194 injected into the abdomen.
  Interventions: Biological: MK-6194
- Thigh Injection (Experimental): Participants will receive a single dose of MK-6194 injected into the thigh.
  Interventions: Biological: MK-6194

INTERVENTIONS:
Biological: MK-6194 — single injected dose
  Other Names: PT101

SUMMARY:
The goal of this study is to learn what happens to MK-6194 in a healthy person's body when different injection sites are used. Researchers will compare what happens to MK-6194 in a healthy person's body when it is injected into the abdomen and when it is injected into the thigh. Researchers think that the average amount of MK-6194 in a person's body over time will be similar when injected into the thigh or abdomen. They also want to learn if it is safe to inject MK-6194 into the abdomen and thigh, and if people tolerate it.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health
* Has a body mass index (BMI) within 18 to 35 kg/m2 and weighs at least 50 kg

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of MK-6194 | At designated timepoints (up to approximately 4 weeks postdose)
  Blood samples will be collected to determine the AUC0-Last of MK-6194.
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of MK-6194 | At designated timepoints (up to approximately 4 weeks postdose)
  Blood samples will be collected to determine the AUC0-Inf of MK-6194.
Maximum Plasma Concentration (Cmax) of MK-6194 | At designated timepoints (up to approximately 4 weeks postdose)
  Blood samples will be collected to determine the Cmax of MK-6194.
Time to Maximum Plasma Concentration (Tmax) of MK-6194 | At designated timepoints (up to approximately 4 weeks postdose)
  Blood samples will be collected to determine the Tmax of MK-6194.
Apparent Clearance (CL/F) of MK-6194 | At designated timepoints (up to approximately 4 weeks postdose)
  Blood samples will be collected to determine the CL/F of MK-6194.
Apparent Terminal Half-life (t1/2) of MK-6194 | At designated timepoints (up to approximately 4 weeks postdose)
  Blood samples will be collected to determine the t1/2 of MK-6194.
Apparent Volume of Distribution (Vz/F) of MK-6194 | At designated timepoints (up to approximately 4 weeks postdose)
  Blood samples will be collected to determine the Vz/F of MK-6194.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event | Up to approximately 12 weeks
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Due to an AE | Up to approximately 12 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- QPS-MRA, LLC-Early Phase (Site 0001), South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com